CLINICAL TRIAL: NCT05816551
Title: Impact of Aging on Gastrointestinal Barrier Function During Hyperthermia
Brief Title: Aging and Gastrointestinal Barrier Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Craig Crandall, Professor, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STU-2023-0171
Record Dates: First submitted 2023-03-15; First posted 2023-04-18 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Aging; Hyperthermia
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Younger participants (Experimental): Individuals aged 18-39 years.
  Interventions: Other: Hyperthermia Trial; Other: Control Trial
- Older participants (Experimental): Individuals aged over 65 years.
  Interventions: Other: Hyperthermia Trial; Other: Control Trial

INTERVENTIONS:
Other: Hyperthermia Trial — Individuals will be exposed to a controlled hyperthermia trial during "Visit 2" of the protocol.
Other: Control Trial — Individuals will be exposed to a control trial (no hyperthermia) during "Visit 1" of the protocol.

SUMMARY:
The purpose of this study is to assess the gastrointestinal responses of the elderly and younger populations during hyperthermia.

DETAILED DESCRIPTION:
Heat waves are lethal and cause a disproportionate number of deaths in the elderly relative to any other age group. Although gastrointestinal barrier dysfunction is a primary cause of heat related illness, little is known about the effects of aging on gastrointestinal barrier function during hyperthermia. The central hypothesis of this work is that the elderly exhibit greater gastrointestinal barrier dysfunction during hyperthermia. Participants will complete a control trial where gastrointestinal permeability (without heating) will be assessed in young and older adults. In the experimental trial, controlled hyperthermia will be achieved using a water perfused, tube lined suit. Core body temperature will be raised to a maximum of 2 degrees Celsius above the baseline value, or an absolute temperature of 39.5 degrees Celsius. Core temperature will not be collected during the control trial. Comprehensive assessments of gastrointestinal barrier function and systemic inflammation will be assessed in young and older adults. The expected outcome of this work will re-shape our understanding of the consequences of aging on gastrointestinal barrier function during heat waves.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female individuals
* 18-35 years or 65+ years of age
* Free of any underlying moderate to serious medical conditions

Exclusion Criteria:

* Known heart disease
* Any chronic medical conditions requiring regular medical therapy including cancer, diabetes, uncontrolled hypertension, inflammatory bowel disease, and uncontrolled hypercholestrolmia etc;
* Abnormality detected on routine screening suggestive of provocable ischemia or previously undetected cardiac disease or resting left bundle branch block on screening electrocardiogram.
* Current smokers, as well as individuals who regularly smoked within the past 3 years
* Subject with a body mass index ≥35 kg/m2
* Pregnant
* Use of immunosuppressant drugs within last 4 weeks prior to screening
* Use of antibiotics or antimicrobial medication in last month
* Any previous abdominal surgery
* Use of steroids in last 6 weeks
* Regular use of probiotics in last month
* Use of laxatives or anti-diarrhetic in last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig G Crandall, Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Texas Health Presbyterian Hospital Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Younger Participants: Individuals aged 18-39 years
  Hyperthermia Trial Individuals will be exposed to a controlled hyperthermia trial during "Visit 2" of the protocol.
  Control Trial Individuals will be exposed to a control trial (no hyperthermia) during "Visit 1" of the protocol.
- Older Participants: Individuals aged over 65 years
  Hyperthermia Trial Individuals will be exposed to a controlled hyperthermia trial during "Visit 2" of the protocol.
  Control Trial Individuals will be exposed to a control trial (no hyperthermia) during "Visit 1" of the protocol.
Period: Overall Study
Arm/Group | Younger Participants | Older Participants
Started | 12 | 10
Control Trial | 11 | 9
Hyperthermia Trial | 12 | 9
Completed (3 participants were withdrawn from the study.) | 9 | 9 (1 participant withdrew from the study.)
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Withdrawn by Primary Investigator | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Younger Participants: Individuals aged 18-39 years
  Hyperthermia Trial: Individuals will be exposed to a controlled hyperthermia trial.
  Control Trial: Individuals will be exposed to a control trial (no hyperthermia).
- Older Participants: Individuals aged over 65 years
  Hyperthermia Trial: Individuals will be exposed to a controlled hyperthermia trial.
  Control Trial: Individuals will be exposed to a control trial (no hyperthermia).
- Total: Total of all reporting groups
Arm/Group | Younger Participants | Older Participants | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 0 | 9
  >=65 years | 0 | 9 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (3) | 72 (3) | 52 (21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 9 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Log Lactulose/Rhamnose Following Control Trial
Description: In vivo gastrointestinal permeability measured by quantities of orally ingested multi-sugar drink excreted in urine. The urinary recovery of each ingested sugar (lactulose, sucrose and rhamnose) was determined by multiplying the measured concentration of each sugar by the total volume of urine collected and dividing by the dose administered. Since lactulose is degraded in the colon, we used the ratio urine lactulose to rhamnose (L/R) to determine small intestinal barrier permeability.
Time Frame: "Visit 1": 3-5 hours after ingestion of multiple sugar drink.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Younger Participants | Older Participants
Number analyzed (Participants) | 9 | 9
Ratio | 0.97 (0.39) | 0.79 (0.30)

2. Primary Outcome: Log Lactulose/Rhamnose Following Hyperthermia Trial
Description: as for outcome 1
Time Frame: "Visit 2": 3-5 hours after ingestion of multiple sugar drink.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Younger Participants | Older Participants
Number analyzed (Participants) | 9 | 9
Ratio | 1.22 (0.32) | 1.21 (0.29)

3. Primary Outcome: Log Sucrose Following Control Trial
Description: The urinary recovery of sucrose was determined by multiplying the measured concentration of sucrose by the total volume of urine collected and dividing by the dose administered. Sucrose is broken down rapidly in the duodenum, thus we used the urinary excretion of sucrose to assess and gastroduodenal permeability.
Time Frame: "Visit 1": 3-5 hours after ingestion of multiple sugar drink.
Measure: Mean (Standard Deviation); unit: log(ng/mL)
Arm/Group | Younger Participants | Older Participants
Number analyzed (Participants) | 9 | 9
log(ng/mL) | 2.68 (1.11) | 1.74 (1.66)

4. Primary Outcome: Log Sucrose Following Hyperthermia Trial
Description: as for outcome 3
Time Frame: "Visit 2": 3-5 hours after ingestion of multiple sugar drink.
Measure: Mean (Standard Deviation); unit: log(ng/mL)
Arm/Group | Younger Participants | Older Participants
Number analyzed (Participants) | 9 | 9
log(ng/mL) | 2.83 (1.10) | 3.44 (0.50)

5. Secondary Outcome: Change in Core Temperature During Hyperthermia Trial
Description: Core temperature was measured using an orally ingestible telemetric pill that was taken no less than 1 hour before the baseline period.
Time Frame: "Visit 2": At 0 minutes and 50-90minutes into the hyperthermia trial.
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Younger Participants | Older Participants
Number analyzed (Participants) | 9 | 9
°C | 2.01 (.14) | 1.95 (.23)

ADVERSE EVENTS:
Time Frame: During the two trials of the experiment or approximately 2 weeks.
Groups:
- Younger Participants Hyperthermia Trial: Individuals aged 18-39 years
  Hyperthermia Trial: Individuals will be exposed to a controlled hyperthermia trial.
- Older Participants Hyperthermia Trial: Individuals aged over 65 years
  Hyperthermia Trial: Individuals will be exposed to a controlled hyperthermia trial.
- Younger Participants Control Trial: Individuals aged 18-39 years
  Control Trial: Individuals will be exposed to a control trial (no hyperthermia).
- Older Participants Control Trial: Individuals aged over 65 years
  Control Trial: Individuals will be exposed to a control trial (no hyperthermia).
Arm/Group | Younger Participants Hyperthermia Trial | Older Participants Hyperthermia Trial | Younger Participants Control Trial | Older Participants Control Trial
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/9 | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9 | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/12 | 1/9 | 0/11 | 0/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Younger Participants Hyperthermia Trial (N=12) | Older Participants Hyperthermia Trial (N=9) | Younger Participants Control Trial (N=11) | Older Participants Control Trial (N=9)
Syncope (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-10-07): https://cdn.clinicaltrials.gov/large-docs/51/NCT05816551/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-07): https://cdn.clinicaltrials.gov/large-docs/51/NCT05816551/SAP_001.pdf